CLINICAL TRIAL: NCT00937612
Title: A Phase II Trial of Postoperative Concurrent Chemoradiation for Head and Neck Squamous Cell Carcinoma Patients With Multiple Risk Factors of Recurrence
Brief Title: Postoperative Concurrent Chemoradiation for Head and Neck Cancer With Multiple Minor Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study group showed better results. Poor Accrual.
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kang-Hsing Fan, Doctor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGHN-0801
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Head and Neck Neoplasms; Carcinoma, Squamous Cell
Keywords: Head and Neck Neoplasms; Chemotherapy; Radiotherapy, Adjuvant; Surgery
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- concurrent chemoradiation (Experimental): patients who has 3 or more minor risk factors of recurrence, and will receive postoperative chemoradiation.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — postoperative radiotherapy, 60-66 Gy/30-33 fractions, concurrently with triweekly chemotherapy by Cisplatin
  Other Names: CGHN 3R trial

SUMMARY:
The purpose of this study is to determine the treatment outcome of postoperative concurrent chemoradiation for head and neck squamous cell carcinoma with multiple minor risks.

DETAILED DESCRIPTION:
Currently, postoperative chemoradiation is recommended for head and neck squamous cell carcinoma with some poor prognostic feature, such as extracapsular spread of metastatic lymph node, or positive resection margin. Other patients may receive postoperative radiotherapy only, if they have other risk factors. In our previous study, if there are 3 or more "minor" risk factors, the 3-year recurrence rate was 55%. This outcome was far inferior to patients who had minor risk factors less than 3. Thus, we believe that current postoperative radiotherapy is insufficient for patients with multiple minor risks. A clinical trial should be raised to help these patients. However, the patient number of this group is not enough for large scale, phase 3 trial. So we arranged this phase II trial of postoperative chemoradiation to test and prospectively observe the treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Primary squamous cell carcinoma of head and neck, after tumor excision and neck dissection, pathology has confirmed three or more of the following adverse prognostic factors, including:

  1. Marginale surgery but a safe distance from the residual tumor ≦ 4mm.
  2. The tumor is located in the hard palate or the retromolar region.
  3. Poorly differentiated cell type.
  4. Tumor invasion to the nerve.
  5. Tumor invasion to lymphatic vessels.
  6. Tumor invasion to the small blood vessels.
  7. Tumor invasion to the bone.
  8. Tumor invasion to the skin.
  9. Depth of tumor invasion ≧ 10mm.
  10. Occurred in single lymph node metastasis.

Exclusion Criteria:

* No or presence of adverse prognostic factor but less than 2.
* Presence of either one conditions listed here: positive resection margin, resection margin negative but less than 1 mm, pathologic N2 or N2, or presence of nodal metastasis with extracapsular spreading.
* ECOG performance status > 2.
* Previous cancer history (except basal cell or squamous cell skin cancer) or other synchronous malignant disease.
* Women during pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2011-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Any kind of cancer recurrence, measured by physical examination or image study. Pathologic confirmation is recommended. | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Kang-Hsing Fan, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (3):
- Taiwan (3):
  - Chang Gung Memorial Hospital, Keelung branch, Keelung
  - Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District
  - Department of Radiation Therapy, Chang Gung Memorial Hospital, Linkou branch, Taoyuan District